CLINICAL TRIAL: NCT06679933
Title: Relationship Between Grip Strength and Intraoperative Hemodynamic Parameters in Geriatric Patients Undergoing Spinal Anesthesia
Brief Title: Relationship Between Grip Strength and Intraoperative Hemodynamic Parameters
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Fatma Nur Arslan, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2021-19/192
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hypotension During Surgery; Geriatric Patient; Hand Grip Strength
Keywords: Geriatric Anesthesia; Hang Grip Strength; Intraoperative Hypotension; Spinal Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Hand grip strength measurament — That intervention includes making the patient sit down and rest for 5 minutes on a comfortable chair. Then make them handle a hand dynamometer with their dominant hand and ask them to squeeze it with all of their effort. Repeat that squeeze three times with 2-minute intervals. The highest number recorded on the dynamometer is the hand grip strength of the patient.

SUMMARY:
In geriatric anesthesia, hand grip strength is used as an important biomarker to evaluate the general health status of elderly patients. Hand grip strength is considered an indicator of various factors, such as muscle function, physical endurance, nutritional status, and frailty, and can be helpful in geriatric anesthesia practice to predict patients' response to anesthesia and determine their risk.

Hand grip strength is used as an important parameter in the pre-anesthesia evaluation of elderly patients. Low grip strength has been associated with postoperative complications (e.g., infection, pulmonary complications, prolonged hospitalization) and worse outcomes.Weak hand grip strength is related to the patient's degree of frailty. Frail patients may be less resistant to stress and respond more negatively to anesthesia.

One of the most important of these responses is intraoperative hypotension, and it is especially common in elderly patients. Since hypotension has possible adverse effects in the postoperative period, it is necessary to evaluate elderly patients in more detail during the preoperative evaluation in order to predict this and take the necessary precautions. Hand grip strength has been found to be associated with cardiovascular system health. With this study, the investigators wanted to evaluate whether measuring hand grip strength during preoperative evaluation would help evaluate the risk of intraoperative hypotension.

DETAILED DESCRIPTION:
One of the most common intraoperative complications following spinal anesthesia is hypotension, which can occur in 16-33% of patients. In non-cardiac surgeries, there is a significant increase in postoperative major cardiac and cerebrovascular events within 30 days, parallel to the decrease in intraoperative mean arterial pressure within hypotensive limits. While there are different threshold values related to mean arterial pressure that can lead to organ damage in the literature, high-quality studies have found this value to be approximately 65 mmHg. However, in elderly patient groups, hypertension is frequently seen due to age-related arterial degeneration, which raises the perfusion thresholds of vital organs. In this context, rather than using a fixed threshold value, the variation of mean arterial pressure may provide a healthier perspective.

The risk of hypotension increases with physiological changes in the elderly, and the more widespread use of spinal anesthesia compared to general anesthesia in older adults underscores the need for better identification of risk factors.

Hand grip strength is a frequently used muscle strength measurement method in sports medicine and geriatric patient groups. It is usually measured in kg or lb with the help of a dynamometer. It provides valuable information in both rehabilitation studies and sarcopenia evaluation. Sarcopenia, or muscle wasting, is associated with frailty in geriatric patients and is one of the important indicators of cardiovascular health. For this reason, the deterioration of cardiovascular health with aging and the increase in the risk of hypotension, one of the side effects of anesthesia, can be predicted by muscle strength evaluation. The aim of our study is to examine whether muscle strength assessment is associated with intraoperative hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 65 years and older
* Patients undergoing elective surgery
* Patients suitable for spinal anesthesia

Exclusion Criteria:

* Presence of anatomical or neurological dysfunction of the upper extremity
* Failed spinal anesthesia
* Failure to measure hand grip strength accurately

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male and female patients over the age of 65 with an ASA score of 1-3 who underwent elective surgery in our hospital (Kırşehir Research and Education Hospital) were included in the study. Patients were selected and included in the study during preoperative evaluation at the anesthesia clinic.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Is low grip strength related with more hypotension? | During the surgery
  We examined whether low hand grip strength was associated with the frequency of intraoperative hypotension.

SECONDARY OUTCOMES:
Is there any difference in blood pressure changes between patients with low hand grip strength and patients with high hand grip strength. | During the surgery
  Male and female participants were evaluated in two separate groups, and a threshold value was determined for hand grip strength in accordance with the literature. The temporal change in blood pressures of patients below and above this threshold value was examined and whether there was a difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Research and Education Hospital, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Gregory A, Stapelfeldt WH, Khanna AK, Smischney NJ, Boero IJ, Chen Q, Stevens M, Shaw AD. Intraoperative Hypotension Is Associated With Adverse Clinical Outcomes After Noncardiac Surgery. Anesth Analg. 2021 Jun 1;132(6):1654-1665. doi: 10.1213/ANE.0000000000005250. PMID 33177322
- [Result] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111